CLINICAL TRIAL: NCT02050425
Title: Exhaled Breath Analysis by Mass Spectrometry in Patients With Obstructive Sleep Apnoea - a Randomised Placebo-controlled Trial.
Brief Title: Breath Analysis in Obstructive Sleep Apnoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Malcolm Kohler, Prof. Dr. med., University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: KEK-2013-0536
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Obstructive Sleep Apnoea (OSA)
Keywords: OSA; CPAP; exhaled breath
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic CPAP (Active Comparator): Patients continue therapeutic continuous positive airway pressure (CPAP).
  Interventions: Device: CPAP
- Subtherapeutic CPAP (Placebo Comparator): Placebo-CPAP device delivering subtherapeutic pressure for two weeks.
  Interventions: Device: Placebo-CPAP device

INTERVENTIONS:
Device: Placebo-CPAP device — short-term CPAP withdrawal by the use of Placebo-CPAP
  Other Names: subtherapeutic CPAP
  Arms: Subtherapeutic CPAP
Device: CPAP — Patients continue therapeutic CPAP therapy
  Arms: Therapeutic CPAP

SUMMARY:
Clinical trial in patients with obstructive sleep apnoea that are randomised to either continue or withdraw continuous positive airway pressure therapy to identify a disease-specific exhaled breath pattern by mass spectrometry.

DETAILED DESCRIPTION:
Randomised placebo-controlled trial (therapeutic vs. subtherapeutic continuous positive airway pressure [CPAP]) including 30 OSA patients to define the effects of CPAP withdrawal (subtherapeutic CPAP) on the composition of exhaled breath analysed by mass spectrometry for identification of OSA specific markers.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed OSA (at the time of original diagnosis) with an oxygen desaturation index (ODI) of >20/h.
* Currently >20/h oxygen desaturations (≥4% dips) during an ambulatory nocturnal pulse oximetry performed on the last night of a 4-night period without CPAP.
* Treated with CPAP for more than 12 months, minimum compliance 4h/night, apnoea-hypopnoea index (AHI) <10 with treatment (according to CPAP- download) and current ESS <10.
* Age between 20 and 75 years at trial entry.

Exclusion Criteria:

* Previous ventilatory failure (awake SpO2 <93% and PaCO2>6kPa).
* Unstable, untreated coronary or peripheral artery disease, severe arterial hypertension or hypotension (>180/110 or <90/60mmHg)
* Previously diagnosed with Cheyne-Stokes breathing.
* Current professional driver; any previous sleep related accident.
* Acute inflammatory disease.
* Acute or chronic hepatic disease.
* Renal failure or renal replacement therapy.
* Use of inhaled drugs.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Exhaled breath pattern. | at baseline and at follow-up (2 weeks)
  OSA-specific mass spectrometric exhaled breath pattern.

SECONDARY OUTCOMES:
apnoea-hypopnoea index (AHI) | at baseline and at follow-up (2 weeks)
  measure of sleep apnoea severity
oxygen desaturation index (ODI), 4% dips | at baseline and at follow-up (2 weeks)
  measure of sleep apnoea severity

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Pulmonology, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Thiel S, Haile SR, Peitzsch M, Schwarz EI, Sievi NA, Kurth S, Beuschlein F, Kohler M, Gaisl T. Endocrine responses during CPAP withdrawal in obstructive sleep apnoea: data from two randomised controlled trials. Thorax. 2019 Nov;74(11):1102-1105. doi: 10.1136/thoraxjnl-2019-213522. Epub 2019 Aug 29. PMID 31467191
- [Derived] Stoberl AS, Schwarz EI, Haile SR, Turnbull CD, Rossi VA, Stradling JR, Kohler M. Night-to-night variability of obstructive sleep apnea. J Sleep Res. 2017 Dec;26(6):782-788. doi: 10.1111/jsr.12558. Epub 2017 May 26. PMID 28548301
- [Derived] Schwarz EI, Martinez-Lozano Sinues P, Bregy L, Gaisl T, Garcia Gomez D, Gaugg MT, Suter Y, Stebler N, Nussbaumer-Ochsner Y, Bloch KE, Stradling JR, Zenobi R, Kohler M. Effects of CPAP therapy withdrawal on exhaled breath pattern in obstructive sleep apnoea. Thorax. 2016 Feb;71(2):110-7. doi: 10.1136/thoraxjnl-2015-207597. Epub 2015 Dec 15. PMID 26671307